CLINICAL TRIAL: NCT02730871
Title: Safety and Efficacy With Twice Daily Brinzolamide 1%/Brimonidine 0.2% (SIMBRINZA®) as an Adjunctive Therapy to Travoprost 0.004%/Timolol 0.5% (DUOTRAV®)
Brief Title: Safety and Efficacy of SIMBRINZA® BID as an Adjunctive to DUOTRAV®
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment Challenges
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GLJ576-P001; 2016-000176-20 (EudraCT Number)
Record Dates: First submitted 2016-03-30; First posted 2016-04-07 (Estimated); Results first posted 2019-05-17 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — brinzolamide; Brimonidine Tartrate; Travoprost; Timolol; Solutions; Duotrav

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Simbrinza + Duotrav (Experimental): Brinzolamide 1%/brimonidine tartrate 0.2% ophthalmic suspension, 1 drop instilled 2 times per day in affected eye(s) (09:00 and 21:00 hrs) plus travoprost 0.004%/timolol 0.5% solution, 1 drop instilled in the affected eye(s) daily in the morning (at 9:00) or in the evening (at 21:00) for 42 days (Treatment Phase)
  Interventions: Drug: Brinzolamide 1%/brimonidine tartrate 0.2% ophthalmic suspension; Drug: Travoprost 0.004%/timolol 0.5% solution
- Vehicle + Duotrav (Placebo Comparator): Brinzolamide/brimonidine vehicle, 1 drop instilled 2 times per day in affected eye(s) (09:00 and 21:00 hrs) plus travoprost 0.004%/timolol 0.5% solution, 1 drop instilled in the affected eye(s) daily in the morning (at 9:00) or in the evening (at 21:00) for 42 days (Treatment Phase)
  Interventions: Drug: Brinzolamide/brimonidine vehicle; Drug: Travoprost 0.004%/timolol 0.5% solution

INTERVENTIONS:
Drug: Brinzolamide 1%/brimonidine tartrate 0.2% ophthalmic suspension
  Other Names: SIMBRINZA® suspension
  Arms: Simbrinza + Duotrav
Drug: Brinzolamide/brimonidine vehicle — Inactive ingredients used as placebo comparator
  Arms: Vehicle + Duotrav
Drug: Travoprost 0.004%/timolol 0.5% solution — 1 drop instilled in the affected eye(s) daily in the morning (at 9:00) or in the evening (at 21:00) for up to 10 days during the Screening/Eligibility Phase and 42 days during the Treatment Phase
  Other Names: DUOTRAV®

SUMMARY:
The purpose of this study is to evaluate the additive intraocular pressure (IOP) lowering effect of Brinzolamide 1%/Brimonidine 0.2% (SIMBRINZA®) dosed twice daily (BID) when added to Travoprost 0.004%/Timolol 0.5% (DUOTRAV®) in subjects with open-angle glaucoma or ocular hypertension.

DETAILED DESCRIPTION:
This study is divided into 2 sequential phases for a total of 5 visits. Phase I of the study is the open-labeled Screening/Eligibility Phase, which includes a Screening Visit followed by 2 Eligibility Visits. Phase II of the study is the randomized, double-masked Treatment Phase, which includes 2 on-therapy visits: Visit 4 (at Week 2) and Visit 5 (Week 6, Exit Visit).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open-angle glaucoma (including pseudoexfoliation or pigment dispersion glaucoma) or ocular hypertension.
* Currently on treatment with Travoprost 0.004%/Timolol 0.5% prescribed as approved in the country, on morning or evening dosing for at least 28 days prior to screening, and in the opinion of the Investigator may benefit from further IOP lowering.
* Mean IOP measurements at both the Eligibility 1 and Eligibility 2 visits, in at least 1 eye (the same eye(s) ≥ 19 and ≤ 28 mmHg at 09:00 while on a Travoprost 0.004%/ Timolol 0.5% solution.
* Able to understand and sign an informed consent form that has been approved by an Institutional Review Board/Ethics Committee.
* Willing and able to attend all study visits.

Exclusion Criteria:

* Women of childbearing potential: not postmenopausal for at least 1 year or less than 6 weeks since sterilization, currently pregnant; have a positive result on the urine pregnancy test at Screening; intend to become pregnant during the study period; breast-feeding; or not in agreement to use adequate birth control methods to prevent pregnancy throughout the study.
* Mean IOP > 28 mmHg at any time point in either eye during the Screening/Eligibility Phase.
* Any form of glaucoma other than open-angle glaucoma or ocular hypertension.
* Severe central visual field loss in either eye.
* Chronic, recurrent or severe inflammatory eye disease in either eye.
* Ocular trauma in either eye within the past 6 months prior to the Screening visit.
* Ocular infection or ocular inflammation in either eye within the past 3 months prior to the Screening visit.
* Retinal degeneration, diabetic retinopathy, or retinal detachment in either eye.
* Best-corrected visual acuity score worse than 55 ETDRS letters (equivalent to approximately 20/80 Snellen, 0.60 logMAR or 0.25 decimal) in either eye.
* Other ocular pathology (including severe dry eye) in either eye that may, in the opinion of the Investigator, preclude the safe administration of any study medication.
* Intraocular surgery in either eye within the past 6 months prior to the Screening visit.
* Ocular laser surgery in either eye within the past 3 months prior to the Screening visit.
* Any other condition including severe illness which would make the subject, in the opinion of the Investigator, unsuitable for the study.
* Asthma, history of asthma, or severe chronic obstructive pulmonary disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2016-06-24 (Actual); Primary Completion 2018-07-13 (Actual); Study Completion 2018-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Assoc Global Trial Director, TM Ophtha, Study Director — Alcon Research
Locations (1):
- Contact Alcon for Locations (Europe, Asia, and Latin America), Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from sites located in Argentina, Australia, Belgium, Chile, Columbia, Germany, Greece, Italy, Malaysia, Poland, Spain, Taiwan, and the United Kingdom.
Pre-assignment Details: Of the 173 enrolled, 39 subjects were exited as screen failures prior to randomization. This reporting group includes all randomized subjects (134).
Period: Overall Study
Arm/Group | Simbrinza + Duotrav | Vehicle + Duotrav
Started (All randomized subjects) | 67 | 67
Full Analysis Set (FAS) (Randomized subjects with a baseline assessment who completed at least 1 scheduled on-therapy visit) | 67 | 67
Safety Analysis Set (All subjects who received a dose of masked investigational product) | 67 | 67
Completed (All subjects who completed the treatment phase whether on study treatment or not) | 61 | 67
Not Completed | 6 | 0
Not completed — Adverse Event | 6 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Simbrinza + Duotrav | Vehicle + Duotrav | Total
Number analyzed (Participants) | 67 | 67 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (13.47) | 65.7 (11.77) | 65.7 (12.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 41 | 73
  Male | 35 | 26 | 61
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 50 | 57 | 107
  Black or African American | 2 | 0 | 2
  Asian | 6 | 7 | 13
  Other | 9 | 3 | 12
Intraocular Pressure (IOP) [Mean (Standard Deviation); unit: mmHg] — IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and reported in millimeters mercury (mmHg).
  mmHg | 21.6 (1.78) | 21.8 (1.90) | 21.7 (1.84)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Diurnal Intraocular Pressure (IOP) (Mean of Changes at 09:00 and 11:00 Time Points) at Week 6
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry. Diurnal IOP change was defined as the average of the two changes from baseline (timepoints 9 AM, 11 AM). A more negative change from baseline indicates a greater improvement, i.e., a reduction of IOP. Only one eye (study eye) was used for the analyses.
Time Frame: Baseline, Week 6
Population: Full Analysis Set. At each time point, only subjects with a value at both baseline and that time point are included in the calculation of change.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Simbrinza + Duotrav | Vehicle + Duotrav
Number analyzed (Participants) | 61 | 67
mmHg | -4.5 (2.69) | -2.4 (3.01)
Statistical Analysis 1: Comparison: Simbrinza + Duotrav vs Vehicle + Duotrav; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = -2.15, 95% CI 2-sided [-2.8 to -1.5], Standard Error of Mean 0.342

2. Secondary Outcome: Mean Diurnal IOP at Week 6
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry. Diurnal IOP was defined as the average of the two time points measured (9 AM, 11 AM). A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). Only one eye (study eye) was used for the analyses.
Time Frame: Week 6
Population: Full Analysis Set with non-missing values
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Simbrinza + Duotrav | Vehicle + Duotrav
Number analyzed (Participants) | 61 | 67
mmHg | 17.1 (2.96) | 19.4 (3.45)
Statistical Analysis 1: Comparison: Simbrinza + Duotrav vs Vehicle + Duotrav; Test type: Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -2.15, 95% CI 2-sided [-2.8 to -1.5], Standard Error of Mean 0.342

3. Secondary Outcome: Mean Percentage Change From Baseline in Diurnal IOP at Week 6
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry. Diurnal IOP percentage change was defined as the average of the two changes from baseline (timepoints 9 AM, 11 AM). A more negative percentage change from baseline indicates a greater improvement, i.e., a reduction of IOP. Only one eye (study eye) was used for the analyses.
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Simbrinza + Duotrav | Vehicle + Duotrav
Number analyzed (Participants) | 61 | 67
percentage change | -20.7 (12.00) | -11.1 (13.86)
Statistical Analysis 1: Comparison: Simbrinza + Duotrav vs Vehicle + Duotrav; Test type: Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -9.98, 95% CI 2-sided [-13.1 to -6.9], Standard Error of Mean 1.572

4. Secondary Outcome: Mean Change From Baseline in IOP (09:00, 11:00) at Week 6
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry. A more negative change from baseline indicates a greater improvement, i.e., a reduction of IOP. Only one eye (study eye) was used for the analyses.
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Simbrinza + Duotrav | Vehicle + Duotrav
Number analyzed (Participants) | 67 | 67
mmHg
  Baseline 9:00 Hr | 22.2 (1.84) | 22.5 (1.80)
  Baseline 11:00 Hr | 21.4 (1.93) | 21.4 (2.26)
  Change from Baseline 9:00 Hr: number analyzed (Participants) | 61 | 67
  Change from Baseline 9:00 Hr | -4.4 (3.07) | -3.2 (3.40)
  Change from Baseline 11:00 Hr: number analyzed (Participants) | 61 | 67
  Change from Baseline 11:00 Hr | -5.4 (2.84) | -2.5 (2.98)
Statistical Analysis 1: Comparison: Simbrinza + Duotrav vs Vehicle + Duotrav; Change from Baseline in IOP at 9:00; Test type: Other; p = 0.022, Repeated measures model; Mean Difference (Final Values) = -1.33, 95% CI 2-sided [-2.5 to -0.2], Standard Error of Mean 0.576
Statistical Analysis 2: Comparison: Simbrinza + Duotrav vs Vehicle + Duotrav; Change from Baseline in IOP at 11:00; Test type: Other; p < 0.001, Repeated measures model; Mean Difference (Final Values) = -2.85, 95% CI 2-sided [-3.9 to -1.9], Standard Error of Mean 0.506

5. Secondary Outcome: Mean Percentage Change From Baseline in IOP (09:00, 11:00) at Week 6
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry. A more negative percentage change from baseline indicates a greater improvement, i.e., a reduction of IOP. Only one eye (study eye) was used for the analyses.
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Simbrinza + Duotrav | Vehicle + Duotrav
Number analyzed (Participants) | 61 | 67
percentage change
  Percent change at 9:00 Hr | -20.2 (13.56) | -14.1 (15.10)
  Percent change at 11:00 Hr | -25.0 (12.73) | -11.7 (13.63)
Statistical Analysis 1: Comparison: Simbrinza + Duotrav vs Vehicle + Duotrav; Percentage Change from Baseline in IOP at 09:00; Test type: Other; p = 0.018, Repeated measures model; Mean Difference (Final Values) = -6.15, 95% CI 2-sided [-11.2 to -1.1], Standard Error of Mean 2.567
Statistical Analysis 2: Comparison: Simbrinza + Duotrav vs Vehicle + Duotrav; Percentage Change from Baseline in IOP at 11:00; Test type: Other; p < 0.001, Repeated measures model; Mean Difference (Final Values) = -13.21, 95% CI 2-sided [-17.8 to -8.6], Standard Error of Mean 2.340

ADVERSE EVENTS:
Time Frame: Baseline through study completion, an average of 42 days
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a subject who is administered a study treatment regardless of whether or not the event has a causal relationship with the treatment. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the study protocol. Includes all subjects who received a dose of masked investigational product (Safety Analysis Set).
Groups:
- Simbrinza + Duotrav: All subjects exposed to brinzolamide 1%/brimonidine tartrate 0.2% ophthalmic suspension plus travoprost 0.004%/timolol 0.5% solution
- Vehicle + Duotrav: All subjects exposed to brinzolamide/brimonidine vehicle plus travoprost 0.004%/timolol 0.5% solution
Arm/Group | Simbrinza + Duotrav | Vehicle + Duotrav
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/67 | 1/67
Other Adverse Events (participants affected / at risk) | 0/67 | 0/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Simbrinza + Duotrav (N=67) | Vehicle + Duotrav (N=67)
Dysuria (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2017-04-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT02730871/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-23): https://cdn.clinicaltrials.gov/large-docs/71/NCT02730871/SAP_001.pdf